CLINICAL TRIAL: NCT06372054
Title: Integration of Omics-based Technologies and Artificial Intelligence to Identify Predictive Risk Models in a Air Force's Pilot Cohort for the Maintenance of Safety, Well-being, Health, and Performance to be Translated to Civil Population
Brief Title: TORNADO-Omics Techniques and Neural Networks for the Development of Predictive Risk Models
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: University of Milan (Other); Italian Air Force (Unknown); A-Tono (Unknown); Ministry of Defense, Italy (Unknown)
Responsible Party: Sponsor
Other Study IDs: TORNADO
Record Dates: First submitted 2024-03-21; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-03

CONDITIONS: Oxidative Injury; Stress Physiological; Discogenic Pain; Cardiovascular Risk Factor; Space Maintenance; Epigenetic Changes; LONGEVITY 1; Neuroplasticity; NGS
Keywords: pilots; air force; epigenetic change; environmental exposure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood, urine, salivae
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High-performance Italian Air Force Pilots: The primary study cohort is represented by "super-healthy" high-performance Italian Air Force Pilots, aged between 26 and 38 years, in active flight service.
  Intervention: not applicable
  Interventions: Other: Biological sample collection
- Italian Air Force ground staff: This cohort of Italian Air Force ground personnel will be used as a control group to compare data from the pilot cohort.
  Interventions: Other: Biological sample collection

INTERVENTIONS:
Other: Biological sample collection — Collection of biological samples (blood, urine, saliva) and clinical data

SUMMARY:
The goal of this observational study is to define a personalized risk model in the super healthy and homogeneous population of Italian Air Force high-performance pilots. This peculiar cohort conducts dynamic activities in an extreme environment, compared to a population of military people not involved in flight activity. The study integrates the analyses of biological samples (urine, blood, and saliva), clinical records, and occupational data collected at different time points and analyzed by omic-based approaches supported by Artificial Intelligence. Data resulting from the study will clarify many etiopathological mechanisms of diseases, allowing the creation of a model of analyses that can be extended to the civilian population and patient cohorts for the potentiation of precision and preventive medicine.

DETAILED DESCRIPTION:
The high-performance pilots of the Italian Air Force are "super healthy" individuals subjected to particular working conditions, as changes in temperature, pressure, gravity, acceleration, exposure to cosmic rays and radiation, which determine psycho-physical adaptation mechanisms to maintain homeostasis. However, this environmental exposure may potentially affect human health, well-being and performance.

The study aims to collect exposure data, clinical, physiological data through biosensors and molecular parameters (at different time point), to be integrated by an Artificial Intelligence algorithm expressly trained to create reliable risk models.

The final outcome will consist of the identification of significant biomarkers of pathological risk, in order to better understand the etiopathological mechanisms of many human diseases and apply early and personalized countermeasures to maintain and empower workers' health status and performance, avoiding clinical symptom presentation.

ELIGIBILITY:
Inclusion Criteria:

* Being part of the Italian Air Force, as in active flight service or ground staff
* Age between 26 and 38 years
* Consent to collect biological samples and use the wearable device to monitor exposure parameters

Exclusion Criteria:

* Age < 25 years and > 39 years
* no signature on informed consent

Ages: 26 Years to 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will consist of high-performance Italian Air Force pilots, compared to Italian Air Force ground staff.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-02-05 (Estimated); Study Completion 2027-02-05 (Estimated)

PRIMARY OUTCOMES:
Assessment of flight-related exposure data and molecular modifications | Through study completion, an average of 3 year
  Collection of information on: i) lifestyle, ii) medical examination, iii) previous trauma, iv) cumulative professional exposure to flying, determination of panel of genes and circulating markers to assess prognostic and predictive factors

SECONDARY OUTCOMES:
Assessment of General Health | Through study completion, an average of 3 year
  Recording of general health condition and work stress by General Health Questionnaire by the Effort-Reward Imbalance Questionnaire (ERI)
Assessment of Sleep Quality | Through study completion, an average of 3 year
  Recording of sleep quality by the Sleeping Quality Questionnaire (SQQ)
Assessment of eating habits | Through study completion, an average of 3 year
  Recording of eating habits by Food Frequency Questionnaire (EPIC)
Creation of reliable AI and disease-based models for personalized medicine | Through study completion, an average of 3 year
  Integration of information obtained from anamnesis, questionnaires, biochemical, genomic, epigenomic, proteomic data with the measurement of heart rate, oxygenation, acceleration, external temperature, presence of ultrasound, infrasound and radiation with artificial intelligence algorithm for the creation of reliable models of disease based on personalized medicine

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Marfia, MD, PhD, Principal Investigator — Fondazione IRCCs Ca' Granda Ospedale MAggiore Policlinico, Italian Air Force; Emanuele Garzia, MD, PhD, Study Chair — Italian Air Force; Marco Locatelli, MD, PhD, Study Chair — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico; Francesco Vestito, PhD, Study Chair — Italian Air Force
Locations (1):
- CeMATA - Joint Center for Aerospace Medicine and Advanced Therapy, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
Subject's data will be collected in completely anonymized form.

REFERENCES:
- [Result] Marfia G, Navone SE, Guarnaccia L, Campanella R, Locatelli M, Miozzo M, Perelli P, Della Morte G, Catamo L, Tondo P, Campanella C, Lucertini M, Ciniglio Appiani G, Landolfi A, Garzia E. Space flight and central nervous system: Friends or enemies? Challenges and opportunities for neuroscience and neuro-oncology. J Neurosci Res. 2022 Sep;100(9):1649-1663. doi: 10.1002/jnr.25066. Epub 2022 Jun 9. PMID 35678198
- [Result] Marfia G, Guarnaccia L, Navone SE, Ampollini A, Balsamo M, Benelli F, Gaudino C, Garzia E, Fratocchi C, Di Murro C, Ligarotti GK, Campanella C, Landolfi A, Perelli P, Locatelli M, Ciniglio Appiani G. Microgravity and the intervertebral disc: The impact of space conditions on the biomechanics of the spine. Front Physiol. 2023 Mar 14;14:1124991. doi: 10.3389/fphys.2023.1124991. eCollection 2023. PMID 36998982